CLINICAL TRIAL: NCT04184388
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Hydrolysed Red Ginseng Extract on Improvement of Cognitive Function
Brief Title: Efficacy and Safety of Hydrolysed Red Ginseng Extract on Improvement of Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IH-CF-HRGE
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Function
Keywords: Hydrolysed Red Ginseng Extract; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolysed Red Ginseng Extract (Experimental): Hydrolysed Red Ginseng extract for 1g/day
  Interventions: Dietary Supplement: Hydrolysed Red Ginseng Extract
- Placebo (Placebo Comparator): Hydrolysed Red Ginseng extract for 0g/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolysed Red Ginseng Extract — once a day for 1 p.o., after breakfast(10 ml/day, Hydrolysed Red Ginseng extract for 1g/day) for 12 week
  Arms: Hydrolysed Red Ginseng Extract
Dietary Supplement: Placebo — once a day for 1 p.o., after breakfast(10 ml/day, Hydrolysed Red Ginseng extract for 0g/day) for 12 week
  Arms: Placebo

SUMMARY:
This study was the evaluate the efficacy and safety of hydrolysed red ginseng extract on the improvement of Cognitive Function

DETAILED DESCRIPTION:
This study was 12 weeks, randomized, double-blind, placebo-controlled human trial to evaluate. 100 subjects participated in hydrolysed red ginseng extract or placebo group. To evaluate the changes in the evaluation items when hydrolysed red ginseng extract was taken 12 weeks compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are at least 60 years of age at screening
* Persons who have Korean Mini-Mental Status Examination(K-MMSE) result in 25-28 points
* Persons who agree to voluntary participation and to comply with the Notice after fully hearing and understanding the details of this human trial

Exclusion Criteria:

* Patients with a past history of treatment with Axis I disorder in SCID(Structured Clinical Interview for DSM-IV) which is a structured clinical interview in the Diagnostic and Statistical Manual of Mental Disorders at Screening or who have been treated within the last 3 years
* Patients with BMI(Body Mass Index)<18.5 kg/m^ or 35 kg/m^≤BMI(Body Mass Index)
* Patients with alcohol abuse or dependence within the last 3 months
* Patients who have clinically significant following severe illness (i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.)
* Patients with a history of clinically significant hypersensitivity to ginseng or red ginseng
* Patients taking medicines, health functional foods or herbal medicines related to the improvement of cognitive function and memory within 1 month before screening
* Patients who ingested ginseng and red ginseng extract's health functional food within 1 month before screening
* Patients who whole blood donation within 1 months before the first ingestion or Component blood donation within 2 weeks
* Patients who participate in another human trial within 3 months
* Those who show the following results in the Laboratory test

  * AST, ALT > 3 times upper limit of the normal range
  * Other significant laboratory test opinion
* Patients who are deemed unsuitable for participating in the human trial due to other reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Visual learning test | 12 weeks
  Visual learning test was measured in baseline and 12 week.
Visual working memory test | 12 weeks
  Visual working memory test was measured in baseline and 12 week.
MoCA-K; Korean Version of the Montreal Cognitive Assessment | 12 weeks
  Korean Version of the Montreal Cognitive Assessment(MoCA-K) was measured in baseline and 12 week. The cognitive function evaluation using the Montreal Cognitive Assessment(MoCA-K) is a total of 8 items, and evaluates cognitive functions such as time / execution power, vocabulary, memory, attention, sentence, abstraction, delayed recall, and orientation.
  Time / execution power's total score is 5 points, vocabulary's total score is 3 points, attention's total score is 3 points, sentence's total score is 3 points, abstraction's total score is 2 points, delayed recall's total score is 5 points, orientation's total score is 6 points. It takes about 10 minutes to complete, and the total score is 30 points and total score make sum score. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.

SECONDARY OUTCOMES:
Auditory continuous performance test | 12 weeks
  Auditory continuous performance test was measured in baseline and 12 week.
Verbal learning test | 12 weeks
  Verbal learning test was measured in baseline and 12 week.
PSS; Perceived stress scale | 12 weeks
  Perceived stress scale(PSS) was measured in baseline and 12 week. It consists of 10 questions. Each question is evaluated from 0 (none) to 4 (very often), and 4 items (4, 5, 7, 8) are scored back and added to the remaining questions. The duration of the last month should be presented before implementation (if the duration is longer, the predictability is lowered).
BDI; Beck Depression Inventory | 12 weeks
  Beck Depression Inventory(BDI) was measured in baseline and 12 week. It consists of 21 items including cognitive, emotional, synchronous, and physical symptoms of depression. The total score ranges from 0~63 points for each question. Beck Depression Inventory(BDI) score is 0 ~ 9 points non-depression, 10 ~ 15 is mild depression, 16 ~ 23 is moderate depression, and 24 ~ 63 is severe depression.
BDNF; Brain-derived neurotrophic factor | 12 weeks
  Brain-derived neurotrophic factor(BDNF)(pg/mL) was measured in baseline and 12 week.
TAS(Total antioxidant status) | 12 weeks
  Total antioxidant status(TAS) was measured in baseline and 12 week.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Department of Psychiatry, Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea